CLINICAL TRIAL: NCT07385066
Title: Effects of Transcranial Direct Current Stimulation (tDCS) Combined With Virtual Reality Versus Conventional Physical Therapy on Brain Activity, Cognitive Function, and Gross Motor Skills in Children With Down Syndrome.
Brief Title: Effects of (tDCS) Combined With Virtual Reality Versus CPT on Brain, Cognitive, and GMS in Children With DS.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2229
Record Dates: First submitted 2026-01-14; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (tDCS + Virtual Reality) (Experimental)
  Interventions: Combination Product: Experimental group (tDCS + Virtual Reality)
- Conventional Physical Therapy (Active Comparator)
  Interventions: Diagnostic Test: Conventional Physical Therapy

INTERVENTIONS:
Diagnostic Test: Conventional Physical Therapy — Participants in the control group will receive standard, evidence-based physical therapy targeting gross motor skills, including exercises for strength, balance and functional mobility
  Arms: Conventional Physical Therapy
Combination Product: Experimental group (tDCS + Virtual Reality) — Participants will receive non-invasive tDCS in combination with interactive, task-oriented VR exercises designed to improve gross motor skills such as balance, standing, walking, and functional mobility. Each session will be supervised by licensed physiotherapists
  Arms: Experimental group (tDCS + Virtual Reality)

SUMMARY:
This randomized controlled trial aims to compare the effects of transcranial direct current stimulation (tDCS) combined with virtual reality-based training versus conventional physical therapy on brain activity, cognitive function, and gross motor skills in children with Down syndrome. Children with Down syndrome commonly exhibit motor and cognitive impairments associated with altered neurodevelopment, which may benefit from neuroplasticity-oriented interventions.

DETAILED DESCRIPTION:
Eligible participants will be randomly allocated into two groups. The experimental group will receive tDCS in combination with virtual reality-based training, while the control group will receive only conventional physical therapy. Interventions will be administered by licensed physiotherapists over a defined treatment period. Gross motor outcomes will be assessed using standardized measures such as the Gross Motor Function Measure (GMFM). Cognitive function will be evaluated using age-appropriate cognitive assessments, and brain activity will be assessed using electroencephalography (EEG), where applicable. Assessments will be conducted at baseline and after completion of the intervention period. The study will adhere to ethical principles, including informed consent from parents or guardians, participant confidentiality, and the right to withdraw at any stage.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years diagnosed with Down syndrome by a pediatrician.
* Compromised gross motor performance in standing, walking, running, or jumping domains of the Gross Motor Function Measure (GMFM).
* Stable medical and neurological status.
* Parental/guardian informed consent and cooperation.
* Documented balance difficulties.
* Ability to follow simple instructions in Urdu or locally spoken language.
* Regular accessibility to the intervention site.

Exclusion Criteria:

* Neurological conditions other than Down syndrome.
* Red flag conditions such as tumors, fractures, metabolic diseases, or dislocations.
* Visual, cardiopulmonary, or severe musculoskeletal impairments requiring surgical management.
* Recent surgery in the past 12 months.
* Seizure history or sensitivity to electrical stimulation.
* Presence of metal implants or hearing aids.
* Tactile or sensory processing issues that prevent participation in therapy.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test | 24 Months
  Assesses functional mobility and walking ability. Time in seconds is recorded for the participant to stand from a chair, walk 3 meters, turn, return, and sit down. Shorter times indicate better mobility.
Raven's Colored Progressive Matrices (RCPM) | 24 Months
  Assesses non-verbal reasoning and general cognitive ability. Scoring is based on the number of correct answers, with higher scores indicating better cognitive function.
Pediatric Balance Scale (PBS) | 24 Months
  Assesses balance and postural control. Comprises 14 items scored from 0 to 4. Total score ranges from 0-56, with higher scores indicating better balance
Caregiver Strain Index (CSI) | 18 Months
  Measures caregiver burden and well-being. Contains 13 items scored 0 (No) or 1 (Yes). Total score ranges 0-13; higher scores indicate greater strain.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No